CLINICAL TRIAL: NCT04191395
Title: Evolution and Treatments of Chronic Inflammatory Systemic Diseases: Implementation of a Hospital Cohort in the Gastroenterology, Dermatology and Rheumatology Departments of the University Hospital of Besançon
Brief Title: Evolution and Treatments of Chronic Inflammatory Systemic Diseases
Acronym: MISTIC
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: P/2019/433
Record Dates: First submitted 2019-12-05; First posted 2019-12-09 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Inflammatory Bowel Diseases; Ulcerative Colitis; Crohn Disease; Arthritis, Rheumatoid; Spondyloarthritis; Psoriatic Arthritis; Psoriasis; Verneuil's Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease; Arthritis, Rheumatoid; Spondylarthritis; Arthritis, Psoriatic; Psoriasis; Hidradenitis Suppurativa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Inflammatory bowel disease
- Chronic inflammatory rheumatic disease
- Chronic inflammatory skin diseases

SUMMARY:
Patients with chronic inflammatory diseases (CID) followed in gastroenterology, dermatology and rheumatology have physiopathological, epidemiological and therapeutic focal points. The pathologies concerned are inflammatory bowel diseases (IBD - Crohn's disease [MC] and ulcerative colitis [RCH]), chronic inflammatory skin diseases (psoriasis or Verneuil's disease) and chronic inflammatory rheumatic diseases (rheumatoid arthritis [RA] and spondyloarthritis [SpA] including psoriatic arthritis [PsA]). Presenting one of these diseases is associated with a higher risk of having a second inflammatory pathology, whether the latter is ophthalmological, dermatological, rheumatological or gastroenterological. An association of extra-articular manifestations is observed in 10 to 30% of patients with SpA, and an association of extra-intestinal manifestations is observed in approximately 30% of patients with IBD. No common database for chronic systemic inflammatory diseases currently exists in France.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated for IBD (MC, UC or indeterminate colitis) in the gastroenterology department of Besançon University Hospital
* Subject meeting the clinical, morphological and histological diagnostic criteria for MC, UC or indeterminate colitis or
* Patients treated for chronic inflammatory rheumatism (RA, SpA, PsA) in the rheumatology department of the University Hospital of Besançon Subject meeting the ACR 2010 classification criteria of RA or modified New York criteria of Ankylosing spondylitis or ASAS criteria of axial or peripheral SpA or CASPAR criteria of PsA or
* Patients treated for chronic inflammatory skin disease (Psoriasis, Verneuil's disease) in the dermatology department of the University Hospital of Besançon

Exclusion Criteria:

* Opposition of the patient
* Patients in emergency situation, persons deprived of their liberty, protected minors or adults.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Inflammatory Bowel Disease, Chronic Inflammatory Skin Diseases or Chronic inflammatory rheumatic disease
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2019-12-11 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of a second inflammatory disease | through study completion (up to 10 years)

CONTACTS AND LOCATIONS:
Overall Officials: Clément Prati, Prof., Principal Investigator — CHU Besançon; Lucine Vuitton, MD, Principal Investigator — CHU Besançon
Locations (1):
- CHU Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No